CLINICAL TRIAL: NCT00680511
Title: Development of a Family-Based Treatment for Adolescent Methamphetamine Use
Acronym: AIMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA021695
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Behavior and Mental Disorders; Methamphetamine Disorders
Keywords: methamphetamine abuse
MeSH Terms: conditions — Behavior; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Family therapy combined with methamphetamine-specific group treatment.
  Interventions: Behavioral: Adolescent Methamphetamine Treament (AMT)
- 2 (Active Comparator): Family Therapy.
  Interventions: Behavioral: Functional Family Therapy (FFT)

INTERVENTIONS:
Behavioral: Adolescent Methamphetamine Treament (AMT) — AMT Group Therapy plus Functional Family Therapy (FFT)
  Arms: 1
Behavioral: Functional Family Therapy (FFT) — FFT
  Arms: 2

SUMMARY:
The AIMS study compares a methamphetamine-specific treatment intervention to a treatment-as-usual Functional Family Therapy (FFT) approach for adolescents ages 15 to 19. Adolescents are assigned to one of two treatment conditions: (1) 16 weeks of FFT designed to strengthen family relationships and develop skills for helping the adolescent avoid drug use; or (2) 16 weeks of a combination of FFT and a methamphetamine-specific intervention involving group and individual therapy sessions; Families are assessed using questionnaires and interviews, and adolescents participate in neuropsychological testing, before, during, and after treatment to provide information about family functioning, the adolescent's drug use, the adolescent's peers, and other factors that may contribute to treatment success. Adolescents also provide urine specimens for drug screening at assessment visits. Through a partnership with Oregon Health and Science University (OHSU), adolescents will participate in functional magnetic resonance imaging appointments at the hospital to examine regional brain blood flow during tasks designed to measure impulsivity and risk-taking behaviors. As a treatment development grant, study investigators will study adolescents' acceptance of and response to the newly developed methamphetamine-specific treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 19 years of age.
* Have at least one parent or parent figure willing to participate.
* Meet DSM-IV diagnostic criteria for drug-abuse or dependence, including a specific meth use disorder.
* Reports meth use on at least 5 of the previous 90 days.
* Have contact with the parent on at least 40% of the past 90 days.
* With their parent be willing to accept randomization to one of the two treatment interventions.
* Be willing to participate in the imaging task in the fMRI pilot study.
* Have basic English competency.
* Have sufficient residential stability to permit probable contact at follow-up.

Exclusion Criteria:

* Evidence of psychotic or organic state of sufficient severity to interfere with understanding of study instruments and procedures.
* Have a medical or psychological condition that would preclude undergoing the fMRI scan.
* Have a sibling who is participating in the study.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Substance Use | 6 months

SECONDARY OUTCOMES:
Engagement and retention of adolescent methamphetamine users. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Holly B. Waldron, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute Center for Family and Adolescent Research, Portland, Oregon, United States